CLINICAL TRIAL: NCT06547086
Title: Rapid Eye Movement Restoration and Enhancement for Sleep-deprived Trauma-adaptation
Acronym: REM-REST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: 2024-0352; HR00112490326 (Other Grant/Funding Number: Department of Defense); A538900 (Other: UW Madison); SMPH/PSYCHIATRY/PSYCHIATRY (Other: UW Madison); Protocol Version 6/12/2025 (Other: UW Madison)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Healthy Volunteers
Keywords: Regular nap taker
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Stimulation followed by no stimulation (Experimental): Phase 2 participants will receive stimulation during their nap at the first visit, and no stimulation during their nap at the second visit.
  Interventions: Device: Transcranial electrical stimulation with Temporal Interference (TES-TI)
- No stimulation followed by stimulation (Experimental): Phase 2 participants will not receive stimulation during their nap at the first visit, and receive stimulation during their nap at the second visit.
  Interventions: Device: Transcranial electrical stimulation with Temporal Interference (TES-TI)

INTERVENTIONS:
Device: Transcranial electrical stimulation with Temporal Interference (TES-TI) — TES-TI uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TES-TI.

SUMMARY:
The goal of this clinical trial is to find out whether stimulating the brain with electrical current during naps can increase certain kinds of brain activity that happen during sleep and lead to improvements in emotional health and stress resilience.

Participants will attend up to 3 study visits, each of which may last up to 4-5 hours. During these visits, participants will wear a high density electroencephalography (hdEEG) cap and take a nap.

DETAILED DESCRIPTION:
This is a single-blind, two-phase study. In the first phase, each participant will be assigned a nap length, a trigger region, a stimulation type (difference frequency, multipolar transcranial electrical stimulation with temporal interference (TES-TI), or phase modulation), and a stimulation start time relative to the appearance of spindles and sawtooth waves in their EEG. These parameters will be varied across and within participants who may undergo multiple naps in order to identify optimal parameters for enhancing REM sleep.

Phase II is a single-blind study comprised of 40 participants. Each participant will undergo two 90-minute naps with possible sham or non-sham stimulation conditions. The naps will be on 2 separate visits to the lab with at least 1 week between visits. Conditions on each visit are randomized and counterbalanced. During each visit, participants will complete both the REST-Q and SSS questionnaires. Full HDEEG will be applied as well as 4-16 stimulation electrodes. Participants will then undergo an emotion regulation task (face task) wherein they are presented with positive, negative, or neutral emotional stimuli. This is followed by a resting EEG recording, then a nap up to 90 minutes in duration. Either sham or non-sham stimuli will be applied at times during the nap period. Upon waking, the same questionnaires and emotion regulation tasks will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-50 years
* Medically healthy
* English-speaking (able to provide consent and complete questionnaires)
* Citizen or holding permanent resident status
* Regular napper (1 or more naps per week)

Exclusion Criteria:

* Any current or past history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions
* History or head trauma resulting in prolonged loss of consciousness; or a history of >3 grade 1 concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines
* Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc)
* History of seizures, diagnosis of epilepsy, histoy of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy or plan to become pregnant in the next 6 months
* Any metal in the body
* Any medical devices or implants (i.e. cardiac pacemaker, medication infusion pump, cochlear implant, vagal nerve stimulator) unless otherwise approved by the responsible MD
* Dental implants containing metal
* Any medication that may alter seizure threshold: ADHD stimulants (Adderall, amphetamine); tricyclic/stypical antidepressants (amitriptyline, doxepine, imipramine, maprotiline, nortriptyline, buproprion); antipsychotics (chlorpromazine, clozapine); bronchodilators (theophylline, aminophylline); antibiotics (fluoroquinolones, imipenem, penicillin, cephalosporins, metronidazole, isoniazid); Antivirals (valacyclovir, ritonavir); OTC antihistamines (diphenhydramine, Benadryl)
* Claustrophobia (a fear of small or closed places)
* Back problems that would prevent lying flat for up to two hours
* Regular night-shift work (second or third shift)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Identify effective TES-TI parameters to trigger spindles | Post nap (up to 90 minutes)
  Researchers will do a power analysis on high density EEG data for spindle frequency (11-15Hz) and see if there is increase in this frequency range during/post stimulation.
Identify effective TES-TI parameters to trigger spindles | Post nap (up to 90 minutes)
  Researchers will do a power analysis on high density EEG data for sawtooth wave frequency (3-5Hz) and see if there is increase in this frequency range during/post stimulation.
Identify effective duration of the nap to maximize TES-TI effect on REM sleep | Post nap (up to 90 minutes)
  Researchers will compare the durations of nap (sleep duration on the EEG) within subjects across their multiple visits, as well as across subjects; correlating this with the stimulation parameters
Change in spindles after effective TES-TI intervention | Post nap (up to 90 minutes)
  Changes in sleep spindle density during sleep as measured by portable EEG device.
Change in sawtooth waves after effective TES-TI intervention | Post nap (up to 90 minutes)
  Researchers will do a power analysis on high density EEG data for sawtooth wave frequency (3-5Hz) and see if there is increase in this frequency range during/post stimulation.
Change in score for vigilance task | Baseline to post-nap (up to 90 minutes)
  The vigilance task is a computerized reaction time task where participants are presented with a fixation point on a computer screen. At random, the fixation point will change appearance at which point the participant is to click a provided button as quickly as possible. The latency response is recorded automatically. Faster responses are indicative of higher vigilance.
Change in sleep quality and mood | Baseline to post-nap (up to 90 minutes)
  Sleep quality and mood will be assessed using the Restorative Sleep Questionnaire (REST-Q), a 9-item questionnaire assessing aspects of restorative sleep. Each item is scored on a 5-point Likert scale, scores range from 9-45. A higher score indicates a more restorative sleep
Change in sleepiness | Baseline to post-nap (up to 90 minutes)
  Sleepiness will be measured using the Stanford Sleepiness Scale (SSS). SSS is a measure of subjective alertness on a 7-point scale. A lower score on the scale indicated higher alertness.
Change in emotion response | Baseline to post-nap (up to 90 minutes)
  Emotional response is measured using an emotional processing task. This task involves viewing a series of emotionally charged images (60 positive, 60 negative, 60 neutral). Participants see a randomized set of these images and are asked to evaluate how pleasant and emotionally arousing each image is on respective 9-point Likert scales
Change in Spectral Power in Sawtooth Wave Frequency (3-5Hz) | Baseline to 4 weeks
Change in minutes scored as REM sleep | Baseline to 4 weeks
  EEG data will be recorded during sleep. The sleep EEG data is separated into stages (REM-NREM). This way, it is known how many minutes they spend in each stage.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Tononi, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No